CLINICAL TRIAL: NCT00719654
Title: Alterations in the Plasma Proteome of Early-Onset Severe Preeclampsia
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Other Study IDs: HR # 17495
Record Dates: First submitted 2008-02-19; First posted 2008-07-22 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; Proteome; Pregnancy
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood plasma and a portion of placenta is retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- EOS-Preeclampsia: Women with symptoms of early-onset preeclampsia
- Normal: Women who do not have symptoms of early-onset preeclampsia

SUMMARY:
The hypothesis of this study is that many plasma proteins are altered in concentration and structure in preeclampsia and the elucidation of these alterations will add to the poorly understood pathophysiology of preeclampsia. In this study we will compare the maternal plasma proteomes of early-onset severe preeclampsia versus healthy controls, compare protein expression and quantification of the maternal plasma proteome at the time of diagnosis of EOS-preeclampsia to the plasma proteome of the same affected subject at 48 hours post delivery and we will verify the placental expression of differentially expressed or post-translationally modified proteins found in the plasma of women with EOS-preeclampsia.

DETAILED DESCRIPTION:
Preeclampsia affects 7-10% of all pregnancies and is directly responsible for 50,000 maternal deaths and 900,000 perinatal deaths each year. Preeclampsia remains unpredictable and incurable except through premature delivery of the fetus. It is essential that a better understanding of preeclampsia is obtained.

Proteomics offers a methodology for identification and quantification of each protein fraction found in human plasma in both disease and health. Since proteins are the basic elements of human biology, it is anticipated that alterations in protein posttranslational modification or total protein expression would be indicative and diagnostic of a disease state. Because proteins are recognized to act as messengers through hormone action, act as enzymes to catalyze important organic reactions and serve as structural components of the human body, they are the most representative of the current state of metabolic and structural activity in both the naive and disease state.

Two groups of patients will be enrolled: (1) Patients with EOS-preeclampsia (N=60) and (2) healthy patients with normal pregnancies (N=240). The patients with EOS-preeclampsia will be matched (1:4) with contemporaneous control patients who are carrying a singleton gestation at a similar gestational age. To measure changes in proteins, we will compare proteins in the blood plasma of women with EOS-preeclampsia before and after pregnancy. We will also compare the blood plasmas of healthy versus EOS-preeclamptic women for differences in plasma proteins. Finally, we will examine the placental RNA of patients with EOS-preeclampsia and healthy patients delivered at 35-37 weeks gestation.

ELIGIBILITY:
Inclusion Criteria:

* 20-34 weeks completed gestational age

Exclusion Criteria:

* Multiple gestation
* Chronic hypertension
* Diabetes
* Lupus
* Tobacco Use

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of women who present to MUSC's Women's Health Clinic prior to their 34th week of pregnancy.
Sampling Method: Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2012-04-09 (Actual); Study Completion 2012-04-09 (Actual)

PRIMARY OUTCOMES:
Blood will be drawn from control patients and EOS-preeclampsia patients to test for differences in proteins between control patients and those with EOS-preeclampsia and differences in the proteins of patients with EOS-preeclampsia before and after birth | Once prior to and once after birth

SECONDARY OUTCOMES:
Placental tissue will be collected from women affected by EOS-preeclampsia. | Once, after birth

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Robinson, MD, Principal Investigator — Medical University of South Carolina; Donna Johnson, Study Chair — Medical University of South Carolina, Obstetrics-Gynecology
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States